CLINICAL TRIAL: NCT00323479
Title: A Multicentre, Open Study Assessing Joint Disorders Under ARIMIDEX® (1mg/Day) as Adjuvant Treatment in Post Menopausal Women With Early Breast Cancer
Brief Title: Arthralgia During Anastrozole Therapy for Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5392L00013; 2005-00-5441-19 EUDRACT number
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-03

CONDITIONS: Early Breast Cancer
Keywords: breast cancer treatment; joint disorders
MeSH Terms: conditions — Breast Neoplasms; Joint Diseases | interventions — Anastrozole

INTERVENTIONS:
Drug: Anastrozole — 1mg/Day oral
  Other Names: ARIMIDEX; ZD1033

SUMMARY:
The purpose of this study is to describe the joint symptoms and structural joint changes under anastrozole as adjuvant treatment in postmenopausal women with early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal woman with a breast cancer and scheduled for an adjuvant treatment with anastrozole
* WHO performance status 0, 1 or 2
* Provision of written informed consent

Exclusion Criteria:

* Recurrence of breast cancer, inflammatory rheumatism
* treatment by chondromodulator, oral glucocorticoid, aromatase inhibitor, anti estrogen, Herceptin
* Diabetes treated by insulin
* Severe renal or hepatic disease
* Known hypersensitivity to anastrozole

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca France Medical Director, MD, Study Director — AstraZeneca
Locations (5):
- France (5):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Poitiers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were included by an investigator-oncologist between 15 June 2006 and 31 December 2007
Pre-assignment Details: Patients were included by an investigator-oncologist who followed them up every 3 months over a period of one year (i.e., 5 visits). An investigator rheumatologist carried out the rheumatological evaluations at inclusion and then every 6 months over a period of one year (i.e., 3 visits)
Groups:
- Anastrozole 1 mg: Anastrozole 1 mg once daily
Period: Overall Study
Arm/Group | Anastrozole 1 mg
Started | 114
Safety Population | 110 (Patients who taken at least one dose of treatment)
Completed | 106 (with at least 1 evaluation for primary efficacy endpoint)
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 3
Not completed — house moving | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anastrozole 1 mg
Number analyzed (Participants) | 106
Age Continuous [Mean (Standard Deviation); unit: year] | 62.87 (6.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Events of Arthralgia
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Anastrozole 1 mg
Number analyzed (Participants) | 106
Participants | 37

2. Secondary Outcome: Functional Index of Cochin at 12 Months in Patients Under Anastrozole.
Description: Functional index of cochin score (from 0 to 90) : sum up of 18 questions on activities involving hands (each question scored from 0 = yes without difficulties (best) to 5 = impossible (worst)) based on 99 patients due to missing values.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Anastrozole 1 mg
Number analyzed (Participants) | 99
Units on scale | 4.32 (9.46)

3. Secondary Outcome: Serum Collagen Degradation Type I - CTX-I at 12 Months in Patients Under Anastrozole
Description: Results are based on 97 patients due to missing values
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Ng/mL
Arm/Group | Anastrozole 1 mg
Number analyzed (Participants) | 97
Ng/mL | 0.5 (0.28)

4. Secondary Outcome: Kellgren and Lawrence Score at 12 Months in Patients Under Anastrozole
Description: X ray evaluation of arthritis in 30 articulations ; each articulation scored from (0 = no arthritis to 4 = severe arthritis) based on 92 patients due to missing values
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Anastrozole 1 mg
Number analyzed (Participants) | 92
Units on scale | 12.66 (13.64)

5. Secondary Outcome: Synovial Membrane Thickness at 12 Months in Patients Under Anastrozole
Description: X ray assessment on hands and wrists based on 99 patients due to missing values
Time Frame: 12 months
Measure: Median (Standard Deviation); unit: millimeter
Arm/Group | Anastrozole 1 mg
Number analyzed (Participants) | 99
millimeter | 1.77 (0.62)

6. Secondary Outcome: Percentage of Participant With Therapeutic Maintenance Under Anastrozole
Description: Treatment compliance. results based on 109 patients due to missing values
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Anastrozole 1 mg
Number analyzed (Participants) | 109
percentage of participants | 80.7

ADVERSE EVENTS:
Description: 110 participants were included in the safety population, those who had taken at least one dose of treatment
Arm/Group | Anastrozole 1 mg
Serious Adverse Events (participants affected / at risk) | 6/110
Other Adverse Events (participants affected / at risk) | 106/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole 1 mg (N=110)
Sudden death unexplained (General disorders) | 1
Lymphangitis (Infections and infestations) | 1
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Calculus urinary bladder (Renal and urinary disorders) | 1
Depression worsened (Psychiatric disorders) | 1
General body pain (General disorders) | 1
Parathyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole 1 mg (N=110)
arthralgia (Musculoskeletal and connective tissue disorders) | 59
hot flush (Vascular disorders) | 35
pain in extremity (Musculoskeletal and connective tissue disorders) | 31
asthenia (General disorders) | 17
back pain (Musculoskeletal and connective tissue disorders) | 14
insomnia (Psychiatric disorders) | 12
headache (Nervous system disorders) | 11
vertigo (Ear and labyrinth disorders) | 8
abdominal pain upper (Gastrointestinal disorders) | 6
nausea (Gastrointestinal disorders) | 10
fatigue (General disorders) | 10
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7
musculosketal pain (Musculoskeletal and connective tissue disorders) | 9
neck pain (Musculoskeletal and connective tissue disorders) | 6
breast fibrosis (Reproductive system and breast disorders) | 7
breast oedema (Reproductive system and breast disorders) | 8
breast pain (Reproductive system and breast disorders) | 8
erythema (Skin and subcutaneous tissue disorders) | 7
lymphoedema (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less